CLINICAL TRIAL: NCT03160963
Title: Optimal Manner of Measuring Power Across the Lifespan
Brief Title: Clinical Power Testing Across Human Lifetime
Status: Completed | Type: Observational
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Joseph Signorile, Professor, University of Miami
Other Study IDs: 20161192
Record Dates: First submitted 2017-05-17; First posted 2017-05-19 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Aged
Keywords: elderly

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Ages 18-29: Power testing 18-29 year old men and women
  Interventions: Other: Power Testing
- Ages 30-39: Power testing 30-39 year old men and women
  Interventions: Other: Power Testing
- Ages 40-49: Power testing 40-49 year old men and women
  Interventions: Other: Power Testing
- Ages 50-59: Power testing 50-59 year old men and women
  Interventions: Other: Power Testing
- Ages 60-69: Power testing 60-69 year old men and women
  Interventions: Other: Power Testing
- Ages 70-79: Power testing 70-79 year old men and women
  Interventions: Other: Power Testing
- Ages 80+: Power testing men and women 80 years of age and above
  Interventions: Other: Power Testing

INTERVENTIONS:
Other: Power Testing — Chair stand, vertical jump, computerized squat

SUMMARY:
We will determine when to transition from the common vertical jump to chair stand depending on age and physical activity levels.

DETAILED DESCRIPTION:
Assessing individuals' power, while it is useful in measuring fitness and performance levels, often requires expensive materials. Vertical jump height has been used to assess peak power output using specific regression equations. The issue with this test, although it is often used with older persons, is that it is not practical or useful in assessing the power output in elderly adults due to possible injury risk and lack of familiarity with providing a maximal jump performance. Power is important for elderly adults; because, higher power output in elderly adults has been shown to highly correlate with overall functionality, the ability to do activities of daily living (ADL), and a reduction in fall probability. A recent study examined the capacity of a regression equation to quantify power in elderly adults using a sit-to-stand test and determined; however, the sit-to-stand lacks the difficulty and exhibits a ceiling effect in younger individuals. Therefore, this study will attempt to determine when to transition from the vertical jump to the sit-to-stand, so that the differences in chronological versus physiological age may be determined during aging, and conversely, during improvements through physical or other interventions.

ELIGIBILITY:
Inclusion Criteria:

* between 18 and 89 years old willing to commit to two days of testing

Exclusion Criteria:

* severe musculoskeletal impairment,
* neurological impairment that would affect balance,
* severe cognitive impairment (Mini-mental 19 or below),
* unstable chronic disease state,
* severe vestibular problems
* severe orthostatic hypotension,
* Simultaneous use of cardiovascular, psychotropic and antidepressant drugs.
* Adults unable to consent
* Prisoners
* Pregnant females

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Men and women 18-100
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2017-01-25 (Actual); Primary Completion 2019-08-15 (Actual); Study Completion 2019-08-15 (Actual)

PRIMARY OUTCOMES:
30 second stand-up test | 5 minutes
  The subject will alternate standing a sitting as many times as possible in the 30 second time frame. Wattage (power) will be computed using the equation by Smith et al., Clin Interventions on Aging, 2010.
Countermovement jump test | 5 minutes
  The subject will begin in a standing position, quickly lower the body to a self-determined angle an reach as high as possible. Jump height will be determined by subtracting the height of the jump from standing reach. The power is computed using the Lewis formula.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph F Signorile, PhD, Principal Investigator — University of Miami
Locations (1):
- Max Orovitz Laboratories, Coral Gables, Florida, United States

IPD SHARING:
Plan to Share IPD: No